CLINICAL TRIAL: NCT05674396
Title: 3-5 FrAction Stereotactic Body Radiation Therapy for Palliation of Head and Neck Squamous Cell Carcinoma: the FAST Phase II Randomized Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0648; NCI-2022-10828 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Palliation (Experimental): Participant will be randomized to standard radiation
  Interventions: Radiation: Traditional Palliation
- Stereotactic body radiotherapy (SBRT) (Experimental): Participants will be randomized to receive (SBRT) Stereotactic body radiotherapy.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Participants will receive radiation as per the schedule discussed with the study doctor.
  Arms: Stereotactic body radiotherapy (SBRT)
Radiation: Traditional Palliation — Participants will receive radiation as per the schedule discussed with the study doctor.
  Arms: Traditional Palliation

SUMMARY:
To learn if it is effective to use advanced radiation treatment techniques (stereotactic radiation or "SBRT") to safely deliver a strong dose of radiation to your tumor in a shorter period of time than would typically be feasible with traditional methods.

DETAILED DESCRIPTION:
Objectives:

* To compare local progression-free survival following palliation with SBRT versus traditional fractionations in patients with HN SCC deemed ineligible for curative-intent treatment.
* To compare pain response, symptom burden, toxicity, local control, progression-free survival, and overall survival between the treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide informed consent
* Histologically confirmed squamous cell carcinoma
* Primary tumor site in the head and neck (includes oral cavity, oropharynx, nasopharynx, hypopharynx, larynx, salivary gland, and cutaneous subsites as well as tumors of unknown primary site)
* Ineligible for curative intent treatment after multidisciplinary evaluation (including evaluation by radiation oncologist and surgeon followed by presentation at multidisciplinary tumor board prior to randomization)
* Prior therapy including radiation, surgery, or systemic therapy is permitted unless further radiation is deemed inappropriate by the enrolling physician
* Metastatic disease is permitted

Exclusion Criteria:

* Contraindications to radiotherapy
* Pregnant or lactating women

5.0 PRE-TREATMENT EVALUATION

* History and physical examination including laryngopharyngoscopy by a radiation oncologist and/or head and neck surgeon within 8 weeks prior to randomization.

  o Clinical examination will include a detailed description of disease target including measurement where feasible to facilitate response assessment
* Documentation of smoking history
* Staging imaging within 12 weeks prior to randomization:

  * Contrast-enhanced CT of the neck and chest or
  * MRI of the neck with CT of the chest or
  * Whole body PET/CT
* Histological confirmation of squamous cell carcinoma
* Pregnancy test for women of child-bearing age, within 2 weeks prior to randomization
* Assessment of all baseline symptoms, using CTCAE version 5.0 within 2 weeks prior to randomization.
* Assessment of baseline pain score (NRS) and analgesic use (non-opioid and opioid)
* Completion of QOL scoring within 2 weeks of randomization
* Informed consents must be obtained prior to any study specific activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
M. D. Anderson Symptom Inventory - Head & Neck (MDASI-HN) Questionnaires | through study completion; an average of 1 year.
  M. D. Anderson Symptom Inventory - Head & Neck (MDASI-HN) score range from 0/10
  (0-symptom has not been present)0 to 10 (10-the symptom was as bad as you can imagine it could be)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Reddy, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org